CLINICAL TRIAL: NCT06555445
Title: Effects of Breathing Exercises With and Without Inspiratory Muscle Training on Dyspnea, Lung Volumes and Lung Capacities in COPD Patients
Brief Title: Effects of Breathing Exercises With and Without Inspiratory Muscle Training in COPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0338
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: COPD
Keywords: Respiratory Muscles; Breathing Exercises; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATHING EXERCISE (Experimental): The participants in group A will be engaging in structured breathing exercises, focusing on the following two techniques Diaphragmatic Breathing and Pursed Lip Breathing
  Interventions: Other: BREATHING EXERCISE
- BREATHING EXERCISE REGIMEN COUPLED WITH BREATHER DEVICE (Active Comparator): Participants will use the BREATHER device daily, performing the routine 5-7 days per week
  Interventions: Other: BREATHING EXERCISE; Other: BREATHING EXERCISE REGIMEN COUPLED WITH BREATHER DEVICE

INTERVENTIONS:
Other: BREATHING EXERCISE — Participants will be guided to adopt a deep breathing practice by emphasizing the use of the diaphragm muscle, thereby minimizing the contribution of accessory muscles during inspiration. This approach fosters the efficiency of respiratory mechanics, aiding in the mitigation of dyspnea symptoms. Participants are directed to undertake these exercises 2-3 times per day, dedicating 15-20 minutes per session, consistently over a period of 2 months. Pursed-Lip Breathing .This technique involves exhaling through semi-closed lips, creating a resistance that helps control the rate of exhalation and, thus, optimizes lung volumes and capacities. This exercise is recommended to be performed similarly to diaphragmatic breathing, 2-3 times daily for 15- 20 minutes per session for a period of 2 months
Other: BREATHING EXERCISE REGIMEN COUPLED WITH BREATHER DEVICE — The resistance on the BREATHER device will be adjusted to match each participant's abilities and progression. The resistance level will be challenging yet manageable, ensuring participant comfort. Each daily session will consist of 15-30 minutes with the BREATHER device and can be split into two shorter sessions if necessary. The total duration of this treatment protocol will span 2 months. The BREATHER device will be employed for both inspiratory and expiratory muscle training. Alongside the device usage, specific breathing exercises, such as diaphragmatic and pursed lip breathing, will be performed
  Arms: BREATHING EXERCISE REGIMEN COUPLED WITH BREATHER DEVICE

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major health issue that affects a large proportion of the population, especially those over 50 years old. It is characterized by breathlessness and reduced lung function. It has been hypothesized that practicing specific breathing exercises could potentially alleviate these symptoms and enhance lung volumes and capacities. In addition, there is a lack of clarity on the effects of inspiratory muscle training along with these breathing exercises, warranting further investigation. To determine the effects of breathing exercises with and without inspiratory muscle training on dyspnea, lung volumes and lung capacities in COPD patients. A total of 46 patients, aged over 50, will be enrolled from National Hospital and medical center, Lahore and Ittefaq Hospital, Lahore. These patients will be randomly divided into two groups A and B: the first group will be assigned to perform only diaphragmatic and pursed lip breathing exercises daily for 2 months. In contrast, the second group will also receive breather, which will involve inhaling through a mouthpiece with variable resistance and using breath-holding techniques. The trial will follow strict ethical guidelines, with all participants providing informed consent. Outcomes will be measured through pulmonary function tests and the Modified Borg Dyspnea Scale. The study will also obtain the necessary approval from the respective ethical committees of the participating institutions. The data will be analyzed in SPSS 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 35 and 50 years (23).
* Be of any gender.
* Have a clinical diagnosis of COPD, severity ranging according to GOLD stages of COPD II to III stages (24).
* Have the functional ability to perform the prescribed breathing exercises and inspiratory muscle training (25).
* Demonstrate a willingness to participate in the study by providing informed consent

Exclusion Criteria:

* Diagnosed musculoskeletal disorders that could potentially interfere with the e execution of the exercises.
* Recent chest injuries that might complicate the respiratory function.
* Pregnancy, given the potential for altered respiratory mechanics and concerns for f fetal safety.
* Prior history of abdominal or pelvic surgeries, as these could affect diaphragmatic movement and overall respiratory function.
* A history of malignancy, due to the potential for compromised overall health status and related complications.
* Active or latent tuberculosis, to prevent exacerbating the condition and potentially spreading the infection.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
6-minute Walk Test (6MWT) | baseline and fourth week
  The 6MWT is a simple and widely used exercise test that measures functional capacity. It provides an objective measure of the patient's ability to perform daily activities and is reflective of submaximal level of functional capacity. In a 6- minute Walk Test (6MWT), the distance covered will depend on the individual's current physical health, age, sex, and other factors. On average, healthy adults may be able to walk between 400 and 700 meters in six minutes. However, individuals with COPD or other respiratory conditions might cover significantly less distance. The test is designed to measure the individual's functional capacity, with the goal being to increase this distance over time through appropriate interventions.
Modified Borg Dyspnea Scale: | baseline and fourth week
  The Modified Borg Dyspnea Scale is a self-reported scale that measures perceived exertion and breathlessness, also known as dyspnea. This scale plays a critical role in assessing how a patient's Chronic Obstructive Pulmonary Disease (COPD) is affecting their quality of life and ability to carry out daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- National Hospital and medical center, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970
- [Background] Worth H, Buhl R, Criee CP, Kardos P, Guckel E, Vogelmeier CF. In 'real world' patients with COPD, exacerbation history, and not blood eosinophils, is the most reliable predictor of future exacerbations. Respir Res. 2023 Jan 5;24(1):2. doi: 10.1186/s12931-023-02311-x. PMID 36604646
- [Background] Kovacs G, Avian A, Bachmaier G, Troester N, Tornyos A, Douschan P, Foris V, Sassmann T, Zeder K, Lindenmann J, Brcic L, Fuchsjaeger M, Agusti A, Olschewski H. Severe Pulmonary Hypertension in COPD: Impact on Survival and Diagnostic Approach. Chest. 2022 Jul;162(1):202-212. doi: 10.1016/j.chest.2022.01.031. Epub 2022 Jan 31. PMID 35092746